CLINICAL TRIAL: NCT03063177
Title: Evaluation of the Associations Between Spinal Manipulative Therapy Dosage and the Related Spinal Stiffness Modulation in Participants With Chronic Thoracic Pain
Brief Title: Evaluation of How Different Dosages of Spinal Manipulation Modulate Spinal Stiffness in Participants With Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, full professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UQTR_2017_dose_stiffness
Record Dates: First submitted 2017-02-20; First posted 2017-02-24 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Back Pain
Keywords: chronic thoracic pain; spine stiffness; spinal manipulation; spinal manipulative therapy
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants won't know the SMT dosage they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1840Newtons/s(N/s);125ms;250 Newtons(N) (Experimental): Participants will receive a spinal manipulative therapy of 20 Newtons (N) preload leading to a peak force of 250N over 125ms (rate of force application of 1840N/s).
  Interventions: Procedure: Spinal manipulative therapy
- 920N/s;125ms;135N (Experimental): Participants will receive a spinal manipulative therapy of 20N preload leading to a peak force of 135N over 125ms (rate of force application of 920N/s).
  Interventions: Procedure: Spinal manipulative therapy
- 920N/s;250ms;250N (Experimental): Participants will receive a spinal manipulative therapy of 20N preload leading to a peak force of 250N over 250ms (rate of force application of 920N/s).
  Interventions: Procedure: Spinal manipulative therapy
- control (No Intervention): Spinal stiffness will be assessed at each sesssion, however, participants won't receive any spinal manipulative therapy.

INTERVENTIONS:
Procedure: Spinal manipulative therapy — A SMT will be delivered by contacting the transverse processes of T7 through our apparatus. Each participant will receive one SMT per session for 3 sessions.
  Arms: 1840Newtons/s(N/s);125ms;250 Newtons(N); 920N/s;125ms;135N; 920N/s;250ms;250N

SUMMARY:
This study evaluate the relationships between spinal manipulative therapy dosage (speed and peak force), the resulting modulation of thoracic spinal stiffness and changes in the clinical status in participants with chronic thoracic pain. Participants will attend four sessions of one hour over 2 weeks. During session 1 to 3, participants will receive one of three different spinal manipulative therapy dosages based on their group assignment and preceded and followed by the measurement of their thoracic spinal stiffness. Session 4 will include spinal stiffness measurement and clinical status evaluation through questionnaires.

DETAILED DESCRIPTION:
Spinal manipulative therapy (SMT) is based on the premise that clinicians can identify spine mechanical changes and accordingly determine the dosage of its biomechanical parameters: preload force, rate of force application and peak force. In recent years, our research team showed, using an apparatus to deliver specific dosage SMTs, that SMT-related neurophysiological responses depend on the dosage of these parameters. Beside determining the SMT dosage, clinicians have to select the spinal level to be treated which is partly done by applying a light pressure to each spinous process (spinal stiffness assessment). This study consist of a randomized controlled trial including 75 participants with chronic thoracic pain who will be randomized in one of three groups. Based on their group assignment, participants will receive a specific dosage SMT delivered at T7 three times over 2 weeks. These SMT dosages are distinct regarding their speed and/or their peak force in order to generate either a high vertebral displacement or a high muscle reflex response. T6, T7 and T8 spinal stiffness will be measured just before and after treatment and clinical status will be assessed at each session beginning through questionnaires. Session four will include the questionnaires and the spinal stiffness measurement procedure. Both SMT and spinal stiffness measurement will be performed using an apparatus aiming at simulating force-time profiles. Surface electromyography electrodes and accelerometers will be positioned over the upper back skin in order to measure the muscle response and vertebral displacement during SMT and spinal stiffness measurement procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 60 years hold and presenting a constant or recurrent pain in the thoracic area for at least 12 weeks. Thoracic are is defined as the region boarded superiorly by T1 spinous process, inferiorly by T12 spinous process and laterally by the lateral border of the thoracic erector spinae muscles. The pain has to be of non organic origin.

Exclusion Criteria:

* Spinal arthritis, aortic aneurysm, collagenosis, advanced osteoporosis, spine surgery, neuromuscular disease, current cancer, uncontrolled hypertension, thoracic radiculopathy, thoracic herniated disc, current infection, thoracic scoliosis, current pregnancy, any contraindication to spinal manipulative therapy of the thoracic spine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Change in spinal stiffness | 2 weeks
  Changes in spinal stiffness between session four and the first session will be assessed at T6, T7 and T8. Spinal stiffness is measured by applying a gradual load of 45 Newtons (N) (5 kg) through our apparatus and by recording the associated indenter displacement. The resulting force-displacement data are used to calculate a spinal stiffness coefficient (N/mm) with lower value indicating more mobility at the spinal level. The change in spinal stiffness will be calculated for each participant by subtracting the value obtained during the fourth session to the one during the first session. A positive value will indicate a decrease in spinal stiffness (increase mobility) while a negative value will indicate an increase in spinal stiffness (decrease mobility) with higher value indicating more important changes.

SECONDARY OUTCOMES:
Change in pain intensity | 2 weeks
  Changes in pain intensity between session four and the first session will be evaluated by subtracting the pain value (over a 0-100 point visual analogue rating scale) obtained at session four by the one at the first session. Positive value indicates a decrease in pain with higher value indicating a more important decrease.

OTHER OUTCOMES:
Change in disability | 2 weeks
  Changes in disability between session four and the first session will be evaluated by subtracting the Quebec Back Pain Disability scale score (0-100 score with higher score indicating higher disability) obtained at session four by the one at the first session. Positive value indicates a decrease in disability with higher value indicating a more important decrease.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, Dc, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Descarreaux M, Nougarou F, Dugas C. Standardization of spinal manipulation therapy in humans: development of a novel device designed to measure dose-response. J Manipulative Physiol Ther. 2013 Feb;36(2):78-83. doi: 10.1016/j.jmpt.2012.12.007. PMID 23499142
- [Derived] Page I, Descarreaux M. Effects of spinal manipulative therapy biomechanical parameters on clinical and biomechanical outcomes of participants with chronic thoracic pain: a randomized controlled experimental trial. BMC Musculoskelet Disord. 2019 Jan 18;20(1):29. doi: 10.1186/s12891-019-2408-4. PMID 30658622